CLINICAL TRIAL: NCT04261894
Title: The OPTIMIZE Study: Optimizing Patient Navigation for Perinatal Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Melissa Simon, Vice Chair of Clinical Research, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SP0052930
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Intervention Model Description: Hybrid Type I Cluster Randomized Effectiveness-Implementation Pragmatic Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OPTIMIZE (Experimental): This arm includes implementation of the OPTIMIZE perinatal care checklist with patient navigation support.
  Interventions: Behavioral: OPTIMIZE
- Standard Care (No Intervention): This arm includes provision of standard perinatal care.

INTERVENTIONS:
Behavioral: OPTIMIZE — The study intervention is implementation of the OPTIMIZE perinatal care checklist with patient navigation support. The checklist will contain perinatal care components to be assessed for each participant. Specifically, the checklist will be built into the electronic health record as a secure digital record of: (1) the participant's adherence to the recommended prenatal and postpartum visit schedule, (2) the completion of procedures and processes in a participant's prenatal and postpartum standard care plan, and (3) the completion of processes to address social determinants of health, along with completion of referrals to appropriate support resources. The OPTIMIZE checklist will also include records of patient navigation review, engagement, and tracking of barrier status and resolution
  Arms: OPTIMIZE

SUMMARY:
This study will develop and test an intervention, called OPTIMIZE, which includes the use of a perinatal checklist by clinic staff and provision of patient navigation support to African American pregnant women. Half of the clinics in the study will be assigned to the OPTIMIZE intervention and half will administer standard care.

DETAILED DESCRIPTION:
African American women and their infants experience profound perinatal health disparities. The purpose of this study is to develop and evaluate the OPTIMIZE intervention, which is an integrated and comprehensive perinatal care checklist with patient navigation support, using a Hybrid Type I Cluster Randomized Effectiveness-Implementation Pragmatic Trial among 600 African American women (15-45 years of age and 1st-2nd trimester of pregnancy) recruited from approximately 20 clinics affiliated with two Chicago area community health center networks that are the largest providers of perinatal care for low-income African American women in Chicago. Clinic sites will be randomized 1:1 to standard perinatal care (control arm) or standard perinatal care plus the OPTIMIZE checklist with Patient Navigation support starting from the initial prenatal visit and up through 12-weeks postpartum (intervention arm).

The study will test the central hypothesis that African American women in the OPTIMIZE intervention group will have received a greater proportion of recommended perinatal care components (prenatal care content, postpartum care content, and social determinants of health content) consistent with American College of Obstetricians and Gynecologists guidelines than African American women in the standard care group.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 to 45 years
* Self-identified as Black/African American
* Pregnant or recently gave birth (less than 6 months post-delivery)
* English speaking

Exclusion Criteria:

* Cognitive impairment
* Incarceration
* Adults unable to consent

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 548 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Receipt of Perinatal Care Components | Baseline through 6 months postpartum
  The primary outcome will be a composite proportion of perinatal care components across three domains, including prenatal care, postpartum care, and social determinants of health content compared between the intervention and control arms.

SECONDARY OUTCOMES:
Rate of breastfeeding | 6 weeks, 3 months, and 6 months postpartum
  Measured by patient report of feedings per day and week
Rate of depressive symptoms | Baseline through 6 months postpartum
  Proportion of women with postpartum depression as measured by Patient Health Questionnaire-9
Rate of postpartum contraception uptake and adherence | Up to 6 months postpartum
  Proportion of women receiving and maintaining contraception
Rate of influenza vaccine uptake | Up to 6 months postpartum
  Proportion of women receiving influenza vaccine
Rate of Tetanus, Diphtheria, Pertussis vaccine uptake | Up to 6 months postpartum
  Proportion of women receiving Tetanus, Diphtheria, Pertussis vaccine
Rate of human papillomavirus vaccine | Up to 6 months postpartum
  Proportion of women receiving human papillomavirus vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Simon, MD, Principal Investigator — Northwestern University
Locations (1):
- ACCESS Community Health Network, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No